CLINICAL TRIAL: NCT03875131
Title: Definition, Quantification, and Utility of Biomarkers of Repetitive Brain Injury in Predicting Concussion and Other Long-Term Injury Risks in Patients With Atrial Fibrillation (Concussion AF)
Acronym: Concussion AF
Status: Completed | Type: Observational
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Other Study IDs: 1050545
Record Dates: First submitted 2019-01-25; First posted 2019-03-14 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Change

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — At each visit a blood sample of 16 mL will be collected for standard blood tests at enrollment, 6,12, 18, and 24 months. Additionally, blood samples will be collected (12 mL) and tested for biomarkers at the time of enrollment, follow-up visits at 6, 12, 18 and 24 months after enrollment. The research staff will keep a portion of the blood that can be used for a future study and it will be maintained in the Intermountain biological specimen repository. Biological samples may be used in current and future research tests multiple times, or until the sample is consumed.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Biomarkers of Dementia and Cognitive Decline — Biomarkers will be obtained at baseline, 6, 12, 18, and 24 months.
  The six questionnaires listed below will be administered at the baseline visit, and repeated at the 24-month visit to evaluate cognitive decline.
  * Mini-Mental Status Evaluation
  * Hachinski Ischemic Scale
  * Cognitive Subscale of Alzheimer's Disease Assessment Scale
  * Disability Assessment for dementia
  * Quality of life improvement as assessed by:
    * Minnesota Living with Heart Failure Scale
    * Anti-Clot Treatment Scale (ACTS) Quality of Life Survey

SUMMARY:
This is a prospective clinical study designed to evaluate biomarkers of brain injury and dementia incidence and moderate cognitive decline rates in moderate- to high-risk atrial fibrillation patients that undergo standard of care atrial fibrillation management.

DETAILED DESCRIPTION:
A written informed consent will be obtained from atrial fibrillation patients seen at Intermountain Medical Center who meet the study eligibility criteria. Following the baseline visit for obtaining informed consent and conduct of baseline procedures, subjects will be required to return to clinic at 6, 12, 18 and 24 months after enrollment. Cognitive testing will be performed at baseline and repeated at 24 months. As much as possible, the study follow-up visits will be scheduled at the same time as the patients' regular visits for clinical care.

Six questionnaires will be administered at the baseline visit and repeated at the 24-month visit. At the time of cognitive assessment, the following will be completed, if not already performed as part of usual standard of care: complete blood count, protime/INR, basic metabolic profile, review of cardiac medications, and review of adverse events and hospitalizations. Additional serum tests will be performed on all subjects at enrollment and at the 24-month visit. Biomarkers will be drawn at specific intervals (baseline, 6, 12, 18, and 24 months) then on an as needed basis (within 7 days) when treatments for atrial fibrillation that may increase brain injury risk occur.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female 65 to ≤ 95 years of age
2. Ability to understand and sign a written informed consent form, which must be obtained prior to initiation of any study procedures
3. AF documented by electrocardiogram, ambulatory event monitor, telemetry, or medical records within 12 months of enrollment
4. Ability to complete a mini-mental status evaluation
5. Ability to independently comprehend and complete a quality of life and dementia questionnaires
6. Willing and able to comply with the follow-up visits, tests, and schedule of evaluations

Exclusion Criteria:

1. Have a history of any form of dementia
2. Have a life expectancy less than 24 months
3. Participation in any other clinical trials involving investigational or marketed products within 30 days prior to entry in the study
4. Other conditions that in the opinion of the Principal Investigator and/or Sub-Investigator(s) may increase risk to the subject and/or compromise the quality of the clinical trial
5. The Principal Investigator and/or Sub-Investigator(s) determine(s) that the subject is not eligible for participation in this research study

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Moderate- to high-risk atrial fibrillation patients that undergo standard of care atrial fibrillation management at Intermountain Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2022-10-24 (Actual); Study Completion 2022-10-24 (Actual)

PRIMARY OUTCOMES:
Incident dementia based on the Mini-Mental Status Examination | 24 months
  For cognitive assessment, the Mini-Mental Status Examination will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.dhs.state.mn.us/main/groups/county_access/documents/pub/dhs16_159601.pdf.
Incident dementia based on the Hachinski Ischemic Scale | 24 months
  For cognitive assessment, the Hachinski Ischemic Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.strokecenter.org/wp-content/uploads/2011/08/hachinski.pdf.
Incident dementia based on the Cognitive Subscale of Alzheimer's Disease Assessment Scale | 24 months
  For cognitive assessment, the Cognitive Subscale of Alzheimer's Disease Assessment Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.adcs.org/Industry/instruments.aspx.
Incident dementia based on the Disability Assessment for Dementia | 24 months
  For cognitive assessment, the Disability Assessment for Dementia will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.statisticssolutions.com/disability-assessment-for-dementia.
Incident dementia based on the Minnesota Living with Heart Failure Scale | 24 months
  For cognitive assessment, the Minnesota Living with Heart Failure Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.queri.research.va.gov/chf/products/hf_toolkit/Minnesota-HF-Questionnaire_Rector.pdf.
Incident dementia based on the Anti-Clot Treatment Scale (ACTS) Quality of Life Survey | 24 months
  For cognitive assessment, the Anti-Clot Treatment Scale (ACTS) Quality of Life Survey will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://hqlo.biomedcentral.com/articles/10.1186/1477-7525-10-120.

SECONDARY OUTCOMES:
Moderate change in cognitive decline based on Mini-Mental Status Examination | 24 months
  For cognitive assessment, the Mini-Mental Status Examination will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.dhs.state.mn.us/main/groups/county_access/documents/pub/dhs16_159601.pdf.
Moderate change in cognitive decline based on Hachinski Ischemic Scale | 24 months
  For cognitive assessment, the Hachinski Ischemic Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.strokecenter.org/wp-content/uploads/2011/08/hachinski.pdf.
Moderate change in cognitive decline based on Cognitive Subscale of Alzheimer's Disease Assessment Scale | 24 months
  For cognitive assessment, the Cognitive Subscale of Alzheimer's Disease Assessment Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.adcs.org/Industry/instruments.aspx.
Moderate change in cognitive decline based on Disability Assessment for Dementia | 24 months
  For cognitive assessment, the Disability Assessment for Dementia will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.statisticssolutions.com/disability-assessment-for-dementia.
Moderate change in cognitive decline based on Minnesota Living with Heart Failure Scale | 24 months
  For cognitive assessment, the Minnesota Living with Heart Failure Scale will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://www.queri.research.va.gov/chf/products/hf_toolkit/Minnesota-HF-Questionnaire_Rector.pdf.
Moderate change in cognitive decline based on Anti-Clot Treatment Scale (ACTS) Quality of Life Survey | 24 months
  For cognitive assessment, the Anti-Clot Treatment Scale (ACTS) Quality of Life Survey will be administered at the baseline visit and repeated at the 24-month visits. More information can be obtained at http://hqlo.biomedcentral.com/articles/10.1186/1477-7525-10-120.

CONTACTS AND LOCATIONS:
Overall Officials: Jared Bunch, MD, Principal Investigator — Intermountain Medical Center
Locations (1):
- Intermountain Medical Center, Murray, Utah, United States

IPD SHARING:
Plan to Share IPD: No